CLINICAL TRIAL: NCT05350215
Title: Effect of Atomoxetine and DAW2022 on OSA Severity
Brief Title: Atomoxetine and DAW2022 on OSA Severity
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Andrew Wellman, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020P002760
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo oral capsules (Placebo Comparator): Placebo (2 pills) before sleep for a week
  Interventions: Drug: Placebo oral capsule
- Atomoxetine and DAW2020 oral capsules (Active Comparator): DAW2020 34 mg 4 h before sleep, single night administration for a week. Simultaneous administration of atomoxetine 40 mg for 3 days 30 min before sleep, 80 mg for the following 4 days, 30 min before sleep
  Interventions: Drug: Atomoxetine Oral Capsule [Strattera]

INTERVENTIONS:
Drug: Placebo oral capsule — Placebo pills for a week, 1 pill 4 hr before sleep and 1 pill 30 min before sleep
  Arms: Placebo oral capsules
Drug: Atomoxetine Oral Capsule [Strattera] — Atomoxetine for a week: 40 mg for 3 days 30 min before sleep, 80 mg for 4 days 30 min before sleep Simultaneous administration of DAW2020 for a week, 34 mg 4 h before sleep
  Other Names: DAW2020 Oral Capsule
  Arms: Atomoxetine and DAW2020 oral capsules

SUMMARY:
Obstructive sleep apnea (OSA) is common and has major health implications but treatment options are limited. In previous research atomoxetine and oxybutynin showed promising effect at reducing OSA severity, however they reduced arousal threshold, one of the key traits responsible for OSA. Since oxybutynin was used mainly as a hypnotic, but it is burdened by several anti-cholinergic side effects, DAW2020, a hypnotic which prolonged the total sleep time in a previous trial in OSA patients, could be a better candidate to associate with atomoxetine.

DETAILED DESCRIPTION:
Two overnight sleep studies will be performed: a drug night and a placebo night, with a month of washout between treatments. The patient will breath spontaneously (without CPAP) for both nights. On the study nights, subjects will present to the laboratory in the evening and be instrumented with a full polysomnography for monitoring sleep, physiological variables (endotypes), and respiratory events. A history and physical examination will be performed on each night prior to beginning the study, as will a urine pregnancy test in premenopausal women. The drugs will be administered as follows. There will be a 3-day run in of atomoxetine 40 mg followed by atomoxetine 80 mg starting on the fourth night until the night of the study. DAW2020 34 mg will be administered for 1-week to allow adequate plasma concentrations to be reached. For the sleep study, at least four hours of sleep (50% in the supine position) will be monitored to assess sleep and respiratory variables.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-to-severe OSA (AHI ≥ 15 events/hr)

Exclusion Criteria:

* All participants will be healthy and without major organ system disease that would preclude undergoing the physiological measurements.
* Use of medications expected to stimulate or depress respiration (including opioids, barbiturates, acetazolamide, doxapram, almitrine, theophylline, 4-hydroxybutanoic acid).
* Use of SNRIs/SSRIs.
* Conditions likely to affect OSA physiology: neuromuscular disease or other major neurological disorder, heart failure (also below), or any other unstable major medical condition.
* Sleep disordered breathing or respiratory disorders other than obstructive sleep apnea:
* Other sleep disorders: periodic limb movements (periodic limb movement arousal index > 10/hr), narcolepsy, or parasomnias.
* Hypersensitivity to the study drug (angioedema or urticaria)
* Contraindications to DAW2020
* Use of medications that lengthen QTc interval
* Hypokaliemia, hypomagnesemia, uncontrolled thyroid disease
* Severe claustrophobia.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Effect of atomoxetine and DAW2020 on OSA severity | 1 week
  OSA severity will be quantified by the number of respiratory events/h (AHI)

SECONDARY OUTCOMES:
Effect of atomoxetine and DAW2020 on arousal index | 1 week
  Arousal index will be calculated as the number of arousal per hour
Effect of atomoxetine and DAW2020 on nadir oxygen desaturation | 1 week
  Nadir oxygen desaturation will be calculated as the lowest oxygen saturation value during sleep

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Messineo L, Preuss M, Azarbarzin A, Vena D, Gell L, Aishah A, Esmaeili N, Kim M, Burdick I, Chen T, White D, Sands SA, Wellman A. Effects of the Combination of Pimavanserin and Atomoxetine on OSA Severity: A Randomized Crossover Trial. Chest. 2025 Jul;168(1):223-235. doi: 10.1016/j.chest.2025.03.013. Epub 2025 Mar 28. PMID 40158847